CLINICAL TRIAL: NCT01353612
Title: Correlation Between Coronary and Carotid Atherosclerotic Disease (CAD) and Links With Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Canadian Atherosclerosis Imaging Network (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAIN-003
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples stored for potential correlation with imaging and cardiovascular outcomes endpoints in subset of patients (optional)
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, multi-center imaging study expecting to enroll approximately 1350 patients scheduled for clinically-indicated coronary angiography. Following informed consent, patient will undergo baseline coronary intravascular ultrasound (IVUS) imaging and non-invasive ultrasound imaging of their carotid arteries. Following a 2-year follow-up period, patients will undergo repeat coronary IVUS and standard invasive coronary angiography as well as carotid ultrasound examination.

Additionally, patients will be contacted by phone on an annual basis for 5 years to collect cardiovascular and cerebrovascular clinical endpoints. Evaluations of plaque burden will be made using invasive and non invasive imaging tools in order to assess correlations between vascular beds, imaging technologies and main cardiovascular events.

DETAILED DESCRIPTION:
CTA and PET Substudy:

A subset of patients enrolled into the main CAIN3 study will undergo a CTA. At sites where both CTA and PET imaging modalities exist, patients will be asked to undergo both tests. The CTA and PET scans can be done separately on 2 imaging beds on different days or performed on the same imaging bed, resulting in a combined CTA and PET scan being done in one scheduled visit. All imaging will be done within 90 days after the follow up IVUS.

The choice of radiotracer used (NaF or FDG) for PET imaging will be dependent upon site and availability on the day of the scan. A total of 120 patients will be enrolled in this substudy with approximately 50-60 undergoing CTA and PET.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 18 years.
* Patients scheduled for clinically indicated coronary angiography and possible ad hoc percutaneous coronary intervention (PCI) will be evaluated before their scheduled procedure.
* Written informed consent (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) obtained prior to any study specific procedures.
* Patients considered to be stable at enrollment (at the discretion of the investigator) are eligible provided they meet all other entry criteria.
* Angiogram meeting qualifying criteria

Exclusion Criteria:

* Women of childbearing potential (women who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who refuse to undergo a urine or serum pregnancy test immediately prior to baseline and repeat imaging evaluations The urine or serum pregnancy test must be negative prior to imaging evaluations.
* Previous coronary artery bypass graft (CABG) surgery or probable need for CABG in the next 24 months.
* Patients who have symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Class III or IV) at baseline.
* Patients with clinically significant valvular heart disease likely to require surgical repair or replacement during the treatment period of the study
* Any clinically significant medical condition or presence of any laboratory abnormality that is considered by the investigator to be clinically important and could interfere with the conduct of the study.
* The presence of severe liver disease as defined by the presence of cirrhosis, chronic active hepatitis, or chronic jaundice with hyperbilirubinemia,
* Patients with eGFR < 45 ml/min prior to baseline imaging procedures, or with nephrotic syndrome
* Patients with a life expectancy less than 2 years.
* History of malignancy (except for curatively treated basal cell or squamous cell carcinoma of the skin) during the 3 years prior to the screening.
* Unable or unwilling to comply with protocol requirements, or deemed by the investigator to be unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical indication for coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 1626 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
co-primary outcome measure - Nominal change from baseline in percent atheroma volume | 2 years
  intravascular ultrasound measure
co-primary outcome measure - nominal change from baseline in carotid IMT | 2 years
  2D B-mode carotid ultrasound measure

SECONDARY OUTCOMES:
cardiovascular morbidity and mortality | 5 years
  as adjudicated by a Clinical Endpoint Committee

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Study Chair — Montreal Heart Institute
Locations (39):
- Canada (39):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Foothills Medical Centre, Calgary, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Interventional Cardiology Research, St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - John Health Science Center, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II - Health Sciences Centre, Halifax, Nova Scotia
  - Cambridge Cardiac Care, Cambridge, Ontario
  - McMaster Clinic Hamilton General Hospital, Hamilton, Ontario
  - St-Mary's Hospital, Kitchener, Ontario
  - KMH Cardiology & Diagnostics Centre, Kitchener, Ontario
  - London Health Sciences Center, London, Ontario
  - KMH Cardiology & Diagnostics Centre, Mississauga, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - Heart Care Research, Oshawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Sunnybrook Health Science Center, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Complexe Hospitalier de la Sagamie, Chicoutimi, Quebec
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - CSSS-Hopital de Gatineau, secteur Hull, Gatineau, Quebec
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - CSSS de Laval, Laval, Quebec
  - Hopital Pierre Boucher, Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM Hopital-Hôtel-Dieu, Montreal, Quebec
  - CUSM Montreal General Hospital, Montreal, Quebec
  - Hopital Sacré-Cœur de Montreal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Centre Hospitalier Régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - Centre de santé et des services sociaux de Beauce, Saint-Georges, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - St. Michael's Hospital, Toronto, Quebec
  - CHRTR de Trois-Rivières, Trois-Rivières, Quebec
  - CSSS Vallée de l'Or, Val-d'Or, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- See also: Canadian Atherosclerosis Imaging Network (CAIN) - "Hearts and Minds" — http://www.canadianimagingnetwork.org/